CLINICAL TRIAL: NCT03850080
Title: Autologous Conditioned Serum: Functional and Clinical Results Using a Novel Disease Modifying Agent for the Management of Knee Osteoarthritis
Brief Title: Autologous Conditioned Serum: Functional and Clinical Results
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Pierluigi Pironti, Doctor, Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1ACS
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Knee Osteoarthritis; Osteoarthritis, Knee; Cartilage Degeneration
Keywords: Knee; Osteoarthritis; Inflammation; Joint; Autologous Conditioned Serum
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Inflammation

STUDY DESIGN:
Intervention Model Description: Single cohort prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Conditioned Serum (Experimental): Patients that were deemed admissible to the trial received 1 intra-articular injection of autologous conditioned serum (Orthokine®) for 4 consecutive weeks at the site of OA. These patients were then followed at 1 month and 6 months for clinical and functional evaluation using VAS for pain, WOMAC, and KSS.
  Interventions: Drug: Autologous Conditioned Serum

INTERVENTIONS:
Drug: Autologous Conditioned Serum — Fifteen patients with clinical and radiological signs of OA of the knee were recruited for this study. 50mL of whole blood were taken using a special syringe containing CrSO4-coated grade glass beads in order to promote IL-1ra synthesis and aggregation.The incubation period lasted 7 hours after which, the blood-filled syringes were centrifuged and the serum supernatant was filtered and aliquoted into four 3mL portions. The aliquots were stored at -20oC until their use was necessary.
  Patients received 1 intra-articular injection for 4 consecutive weeks at the site of OA.
  Other Names: ACS; Orthokine®

SUMMARY:
The purpose of this study was to investigate the potential ability of autologous conditioned serum (ACS) to decrease the pain and improve the joint functionality in patients affected by knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Fifteen patients with clinical and radiological signs of OA of the hip or knee were recruited for this study. Each patient received 4 injections of ACS (Orthokine®) at the site of OA once per week for 4 weeks. Clinical and functional evaluation were performed using VAS scale for pain, WOMAC scale and KSS functional and clinical scores before the first injection, at one week, at two weeks, at three weeks, at one month and at six months. Statistical analysis was done with the Wilcoxon Signed-Rank Test.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis >3 months in clinical and radiographic signs
* VAS for pain >50mm

Exclusion Criteria:

* Hepatitis B
* Hepatitis C
* HIV
* pregnancy
* drug abuse
* other intra-articular injections <6 months
* surgery on affected knee <12 months

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) | 6 months
  24 questions each scaled out of 100mm. 5 questions regarding pain. 2 questions regarding rigidity. 17 questions regarding difficulty in various activities. Total score out of 240 expressed as a percentage. Minimum score 0. Max score 100. Greater score implies worsening symptomatology.
Knee Society Score (KSS) | 6 months
  Clinical Score. Pain is measured out of 50 (no pain = 50, severe pain = 0). Range of motion (1 point for every 5 degress of flexion. Max points = 25). Stability; anteroposterior (<5 degrees 10, 5-10 degrees 5, >10 degrees 0); mediolateral (<5 degrees = 10, 5-10 degrees = 5, >10 degrees = 0); Flexion contracture (5-10 degrees = -2, 10-15 degrees = -5, 16-20 degrees = -10, >20 degrees = -15); Extension lag (<10 degrees = -5, 10-20 degrees = -10, 20 degrees = -15); Alignment (0-4 degrees = 0, 5-15 degrees = 3 points for each degree).
  Functional Score. Consists of walking score based on how many blocks (100m) patient can walk without stopping (unlimited = 100, >10 blocks = 40, 5-10 blocks = 30, <5 blocks = 20, housebound = 10, unable = 0); Stairs (normal = 50, normal up down with support = 40, up and down with support = 30, up with support down unable = 15, unable = 0); Functional deductions (cane = -5, two canes = -10, crutches or walker = -20)
Visual Analog Score for Pain | 6 months
  Subjective evaluation of pain reported by each patient on average since the last visit. Minimum = 0. Maximum = 10

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Vitali, MD, Study Director — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shewale AR, Barnes CL, Fischbach LA, Ounpraseuth ST, Painter JT, Martin BC. Comparative Effectiveness of Intra-Articular Hyaluronic Acid and Corticosteroid Injections on the Time to Surgical Knee Procedures. J Arthroplasty. 2017 Dec;32(12):3591-3597.e24. doi: 10.1016/j.arth.2017.07.007. Epub 2017 Jul 14. PMID 28781020
- [Background] Klocke R, Levasseur K, Kitas GD, Smith JP, Hirsch G. Cartilage turnover and intra-articular corticosteroid injections in knee osteoarthritis. Rheumatol Int. 2018 Mar;38(3):455-459. doi: 10.1007/s00296-018-3988-2. Epub 2018 Feb 2. PMID 29396701
- [Background] Bhandari M, Bannuru RR, Babins EM, Martel-Pelletier J, Khan M, Raynauld JP, Frankovich R, Mcleod D, Devji T, Phillips M, Schemitsch EH, Pelletier JP. Intra-articular hyaluronic acid in the treatment of knee osteoarthritis: a Canadian evidence-based perspective. Ther Adv Musculoskelet Dis. 2017 Sep;9(9):231-246. doi: 10.1177/1759720X17729641. Epub 2017 Sep 12. PMID 28932293
- [Background] Pelletier JP, Martel-Pelletier J, Abramson SB. Osteoarthritis, an inflammatory disease: potential implication for the selection of new therapeutic targets. Arthritis Rheum. 2001 Jun;44(6):1237-47. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-F. No abstract available. PMID 11407681
- [Background] Nuki G. Osteoarthritis: a problem of joint failure. Z Rheumatol. 1999 Jun;58(3):142-7. doi: 10.1007/s003930050164. PMID 10441841
- [Background] Kapoor M, Martel-Pelletier J, Lajeunesse D, Pelletier JP, Fahmi H. Role of proinflammatory cytokines in the pathophysiology of osteoarthritis. Nat Rev Rheumatol. 2011 Jan;7(1):33-42. doi: 10.1038/nrrheum.2010.196. Epub 2010 Nov 30. PMID 21119608
- [Background] Martel-Pelletier J, Alaaeddine N, Pelletier JP. Cytokines and their role in the pathophysiology of osteoarthritis. Front Biosci. 1999 Oct 15;4:D694-703. doi: 10.2741/martel. PMID 10525480
- [Background] Nixon AJ, Grol MW, Lang HM, Ruan MZC, Stone A, Begum L, Chen Y, Dawson B, Gannon F, Plutizki S, Lee BHL, Guse K. Disease-Modifying Osteoarthritis Treatment With Interleukin-1 Receptor Antagonist Gene Therapy in Small and Large Animal Models. Arthritis Rheumatol. 2018 Nov;70(11):1757-1768. doi: 10.1002/art.40668. Epub 2018 Sep 10. PMID 30044894
- [Background] Calich AL, Domiciano DS, Fuller R. Osteoarthritis: can anti-cytokine therapy play a role in treatment? Clin Rheumatol. 2010 May;29(5):451-5. doi: 10.1007/s10067-009-1352-3. Epub 2010 Jan 27. PMID 20108016
- [Background] Alvarez-Camino JC, Vazquez-Delgado E, Gay-Escoda C. Use of autologous conditioned serum (Orthokine) for the treatment of the degenerative osteoarthritis of the temporomandibular joint. Review of the literature. Med Oral Patol Oral Cir Bucal. 2013 May 1;18(3):e433-8. doi: 10.4317/medoral.18373. PMID 23524415
- [Background] Buckland-Wright C. Subchondral bone changes in hand and knee osteoarthritis detected by radiography. Osteoarthritis Cartilage. 2004;12 Suppl A:S10-9. doi: 10.1016/j.joca.2003.09.007. PMID 14698636
- [Result] Baltzer AW, Moser C, Jansen SA, Krauspe R. Autologous conditioned serum (Orthokine) is an effective treatment for knee osteoarthritis. Osteoarthritis Cartilage. 2009 Feb;17(2):152-60. doi: 10.1016/j.joca.2008.06.014. Epub 2008 Jul 31. PMID 18674932
- [Result] Fox BA, Stephens MM. Treatment of knee osteoarthritis with Orthokine-derived autologous conditioned serum. Expert Rev Clin Immunol. 2010 May;6(3):335-45. doi: 10.1586/eci.10.17. PMID 20441419
- [Result] Wehling P, Moser C, Frisbie D, McIlwraith CW, Kawcak CE, Krauspe R, Reinecke JA. Autologous conditioned serum in the treatment of orthopedic diseases: the orthokine therapy. BioDrugs. 2007;21(5):323-32. doi: 10.2165/00063030-200721050-00004. PMID 17896838
- [Result] Auw Yang KG, Raijmakers NJ, van Arkel ER, Caron JJ, Rijk PC, Willems WJ, Zijl JA, Verbout AJ, Dhert WJ, Saris DB. Autologous interleukin-1 receptor antagonist improves function and symptoms in osteoarthritis when compared to placebo in a prospective randomized controlled trial. Osteoarthritis Cartilage. 2008 Apr;16(4):498-505. doi: 10.1016/j.joca.2007.07.008. Epub 2007 Sep 6. PMID 17825587